CLINICAL TRIAL: NCT00642343
Title: Balance in Children With Cochlear Implants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Wayne Berryhill, M.D., University of Oklahoma Health Sciences Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BALANCE W/COCHLEAR_BERRYHILL
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Severe, Profound Deafness
Keywords: Balance; Severe, Profound deafness; Children; unilateral/bilateral cochlear implants; unilateral cochlear implant; bilateral cochlear implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Children with severe to profound deafness that have not received any intervention.
  Interventions: Behavioral: Evaluation of motor proficiency.
- 2 (Active Comparator): Children with an unilateral cochlear implant.
  Interventions: Behavioral: Evaluation of motor proficiency skills.
- 3 (Active Comparator): Children with bilateral cochlear implants.
  Interventions: Behavioral: Evaluation of motor proficiency
- 4 (Active Comparator): Children who receive their second implant during the duration of the study.
  Interventions: Behavioral: Evaluation of motor proficiency

INTERVENTIONS:
Behavioral: Evaluation of motor proficiency skills. — The balance subtest of the Bruininks-Oseretsky Test 2nd Ed. will be administered and scored.
  Other Names: deaf children, balance, unilateral cochlear implants,; bilateral cochlear implants
  Arms: 2
Behavioral: Evaluation of motor proficiency — The balance subtest of the Bruininks-Oseretsky Test 2nd Ed. will be administered and scored.
  Other Names: balance,unilateral/bilateral cochlear implants,; deaf children
  Arms: 3
Behavioral: Evaluation of motor proficiency — The balance subtest of the Bruininks-Oseretsky Test 2nd Ed. will be administered and scored.
  Other Names: balance, unilateral/bilateral cochlear implants,; deaf children
  Arms: 4
Behavioral: Evaluation of motor proficiency. — The balance subtest of the Bruininks-Oseretsky Test 2nd Ed. will be administered and scored.
  Other Names: deaf children, unilateral/bilateral cochlear implants,; balance
  Arms: 1

SUMMARY:
The purpose is to test the balance of children with unilateral,bilateral cochlear implants and patients having unilateral implants before,bilateral implants after surgery,using the Bruininks-Oseretsky Test 2nd ed. to find out if the cochlear implants have an effect.

DETAILED DESCRIPTION:
Hearing impairment has a significant impact on individual quality of life and stresses community resources. In the last two decades cochlear implantation has developed into the new standard of care for severe to profound haring loss. Recent studies have shown bilateral implantation improves sound localization and understanding of speech in noise. For children, this is seen as a significant benefit. As we begin to offer bilateral cochlear implants to a growing number of children it would be in our patient's best interest to evaluate whether or not this may cause balance impairment. We will evaluate the balance scores of children with bilateral cochlear implants, and compare their results to unilaterally implanted children and a hearing impaired population, with the Bruininks-Oseretsky Test 2nd ed (BOT2). In addition we will take a small group of unilaterally implanted patients and test them before and after a contralateral cochlear implant as a prospective study group.

ELIGIBILITY:
Inclusion Criteria:

* Children with cochlear implant(s) activated for at least two weeks before participation.
* Children with severe to profound deafness that have not received intervention.

Exclusion Criteria:

* Children with mental retardation, associated physical handicaps, or chronic sedative use prohibiting completion of the balance tests.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The specific aim will be to compare the balance of children with cochlear implants to profoundly deaf children using the BOT2. | no earlier than 2 weeks following activation of implants

SECONDARY OUTCOMES:
To evaluate the differences in balance function between children with bilateral cochlear implants compared to children with unilateral cochlear using implants the BOT2. | no earlier than 2 weeks after implant activation

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Berryhill, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States